CLINICAL TRIAL: NCT03361904
Title: Adenoma and Advanced Neoplasia Detection Rates Increase From 45 Year of Age: Results of a Monocentric One-year Observational Cohort Study on 6027 Colonoscopies
Brief Title: Colonoscopic Adenoma and Advanced Neoplasia Detection Rates According to Age
Status: Completed | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, KARSENTI, principal investigator, Société Française d'Endoscopie Digestive
Other Study IDs: 2016-ADR according to age
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Colonic Polyp; Colon Adenoma; Colonoscopy; Colon Cancer; Age
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colonoscopy — Total colonoscopy : All consecutive patients who were scheduled for colonoscopy were included. Exclusion criteria were: patients scheduled for partial colonoscopy, interventional colonoscopy (for stent insertion, stenosis dilation).

SUMMARY:
Current recommendations for colonoscopy screening programs usually involve patients older than 50 years of age. However, little is known about polyp or adenoma detection rates under 50. We compared these detection rates according to age in a large series of patients in common practice.

Methods: All colonoscopies performed in 2016 in our unit were prospectively recorded. We determined adenoma detection rate (ADR), polyp detection rate (PDR), mean number of polyps (MNP), and advanced neoplasia detection rate (ANDR).

DETAILED DESCRIPTION:
Patients All consecutive patients who were scheduled for colonoscopy were included. Exclusion criteria were: patients scheduled for partial colonoscopy, interventional colonoscopy (for stent insertion, stenosis dilation).

Data collection The following data have been prospectively collected: age, gender, indication for colonoscopy, preparation procedure and quality of the preparation (assessed by the Boston Bowel Preparation Scale; BBPS) [19-20], caecal intubation (yes/no), withdrawal time, number and size of polyps and polyp histopathology.

All clinical data were collected during the procedure by a nurse and an endoscopist on a dedicated software. The database was then supplemented by the Clinical Research Associate for histopathological data.

We determined adenoma detection rate (ADR; percentage of colonoscopies with at least one adenoma), polyp detection rate (PDR: percentage of colonoscopies with at least one polyp), mean number of polyps per colonoscopy (MNP), large polyp detection rate (LPDR; percentage of colonoscopies with at least one polyp of 1 cm or more) and advanced neoplasia detection rate (ANDR: percentage of colonoscopies with at least one advanced neoplastic lesion as defined below).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who were scheduled for colonoscopy were included.

Exclusion Criteria:

* patients scheduled for partial colonoscopy, interventional colonoscopy (for stent insertion, stenosis dilation).

Ages: 15 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: During the study period, 6335 colorectal endoscopic procedures were realized in the endoscopy unit. We excluded 278 sigmoidoscopies and 30 interventional procedures for stent insertion or stenosis dilation. Only diagnostic colonoscopies were recorded, performed in 3308 women (54.9%) and 2719 men (45.1%) with a median age of 57 (range, 15-96: IQR 18).
Sampling Method: Non-Probability Sample
Enrollment: 6027 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate according to age | during colonoscopy
  ADR <30yo, in 30-34 yo, in 35-39yo, in 40-44yo, in 45-49yo, in 50-54yo, in 55-59yo, in 60-64yo, in 65-69 yo, in 70-74yo, in 75-79yo and >79yo intervals
Advanced Neoplasia Detection rate according to age | during colonoscopy
  ANDR <30yo, in 30-34 yo, in 35-39yo, in 40-44yo, in 45-49yo, in 50-54yo, in 55-59yo, in 60-64yo, in 65-69 yo, in 70-74yo, in 75-79yo and >79yo intervals

SECONDARY OUTCOMES:
Age | during colonoscopy
  years old
Gender | during colonoscopy
  Male or Female
Indication for colonoscopy | during colonoscopy
  pain / screening/ familial or personal history of polyp or cancer
quality of the preparation | during colonoscopy
  Boston Bowel Preparation Scale Segment Score Description 0: unprepared colon segment with mucosa not senn due to solid stool that cannot be cleared
  1. Portion of mucosa of the colon segment seen, but other areas of the colon segment are not well seen due to staining, residual stool, and/or opaque liquid
  2. minor amount of residual staining, small fragments of stool, and/or opaque liquid, but mucosa of colon segments is seen well
  3. entire mucosa of colon segment seen well, with no residual staining, small fragments of stool or opaque liquid
  Total score is a summation of scores from three segments of the colon Score is from 0 to 9
Caecal intubation | during colonoscopy
  Y/N
Withdrawal time | during colonoscopy
  in seconds

CONTACTS AND LOCATIONS:
Overall Officials: David Karsenti, MD, Principal Investigator — Pole Digestif Paris-Bercy

IPD SHARING:
Plan to Share IPD: No